CLINICAL TRIAL: NCT03751787
Title: Interest of Treatment With Cranial Osteopathy in Functional Disorders of the Newborn
Brief Title: Cranial Osteopathy in Functional Disorders of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2008_43; 2009-A00037-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Newborn Complication
Keywords: osteopathy; cranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cranial osteopathy (Experimental): The group will receive treatment with osteopathic cranial osteopathy
  Interventions: Other: cranial osteopathy
- comfort massage (Placebo Comparator): The group will benefit from a placebo manipulation by an osteopathic student who has not yet been trained in cranial osteopathy.
  Interventions: Other: comfort massage

INTERVENTIONS:
Other: cranial osteopathy — two sessions at three weeks intervals
  Arms: cranial osteopathy
Other: comfort massage — manipulation, comfort massage, standardized and not affecting the skull
  Arms: comfort massage

SUMMARY:
To evaluate, from the maternity stay, the interest of the cranial osteopathy in the reduction of the hyper irritability of the newborn and the improvement of the postural abnormalities

ELIGIBILITY:
Inclusion Criteria:

* Newborns:

  * forward
  * born vaginally or cesarean section
  * with or without general anesthesia
  * with or without epidural or spinal anesthesia
  * with or without instrumental extraction
  * presenting at least 1 of the 4 criteria detailed above, numbered at 3 or 4 or two criteria at 2

Exclusion Criteria:

* Newborns presenting:

  * a score of Amiel <7, signing a strong suspicion of non-integrity of brain functions (see table) and therefore leaving the framework of functional pathology
  * symptomatic maternal-fetal infection
  * true obstetric trauma: brachial plexus paralysis, fracture
  * or of a mother who has taken during pregnancy drugs or toxic drugs that affect the behavior of the newborn. (benzodiazepines, subutex, methadone, cocaine, heroin or cannabis)

Ages: 1 Minute to 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction of hyper irritability | at 28 days of life.
  Reduction of hyper irritability will be done by evaluation from a clinical score,signs of hyper irritability during stay in maternity or postural disorders: one of the following 4 criteria rated 3 or 4, or at least two of these rated criteria 2:
  * Excessive and difficult to calm, insufficient sleep
  * postural asymmetry
  * difficulties in feeding, ineffective suckling, including asymmetries (babies breastfeeding and refusing each other), difficulty suckling
  * Excessive regurgitation

SECONDARY OUTCOMES:
Reduction of hyper irritability | before any treatment, at 3 days after deliverance and at 28 days of life
  Reduction of hyper irritability will be done by evaluation from a clinical score, signs of hyper irritability during stay in maternity or postural disorders: one of the following 4 criteria rated 3 or 4, or at least two of these rated criteria 2:
  * Excessive and difficult to calm, insufficient sleep
  * postural asymmetry
  * difficulties in feeding, ineffective suckling, including asymmetries (babies breastfeeding and refusing each other), difficulty suckling
  * Excessive regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Boez, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Maternité Paul Gelé du CH de Roubaix, Roubaix, France

IPD SHARING:
Plan to Share IPD: No